CLINICAL TRIAL: NCT07129733
Title: Oral Care Layered Enhancement for Improved Oral Hygiene in Intensive Care Units: A Stepped-Wedge Cluster Randomized Clinical Trial
Brief Title: Oral Care Layered Enhancement for Improved Oral Hygiene in Intensive Care Units
Acronym: ORACLE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital do Coracao (Other)
Collaborators: Faculdade de Medicina de Ribeirão Preto/USP (Unknown)
Responsible Party: Principal Investigator, Bruno Martins Tomazini, MD, Hospital do Coracao
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: ip_hcor_oracle
Record Dates: First submitted 2025-05-28; First posted 2025-08-19 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: Mechanical Ventilation; Infection Prevention; Oral Care; Oral Hygiene, Oral Health; VAP - Ventilator Associated Pneumonia
Keywords: Oral care; Oral hygiene; critically ill; mechanical ventilation
MeSH Terms: conditions — Pneumonia, Ventilator-Associated; Critical Illness

STUDY DESIGN:
Intervention Model Description: This is a stepped wedge cluster randomized clinical trial, with a 11-month transition period between interventions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Oral hygiene bundle (Experimental): This arm will receive the standardized oral hygiene bundle
  Interventions: Other: Oral hygiene bundle
- Standard of care (No Intervention): Each center will maintain its usual oral care practices.

INTERVENTIONS:
Other: Oral hygiene bundle — Implementation of the standardized oral hygiene bundle, which consists of the following key components: Standardization of materials used during the oral hygiene procedure, standardization of oral hygiene frequency, training of nursing staff involved in patient care on proper oral hygiene practices, discontinuation of routine application of chlorhexidine oral solution, and implementation of a standardized oral hygiene technique.
  Arms: Oral hygiene bundle

SUMMARY:
The goal of the ORACLE study is to evaluate the impact of implementing a standardized oral hygiene bundle on outcomes in critically ill, mechanically ventilated patients. The primary objective is to determine whether this bundle can increase the number of ventilator-free days compared to the standard of care.

DETAILED DESCRIPTION:
The use of invasive mechanical ventilation (IMV) as an organ support measure is common in intensive care units (ICUs), with its prevalence ranging from 36% to 89%. Lower respiratory tract infections (LRTIs) are known to be the primary site of infection related to sepsis in critically ill patients in Brazilian ICUs and are associated with high morbidity and mortality.

It is well established that the oral cavity is a source of pathogens leading to LRTIs in critically ill patients, with dental plaque serving as an important reservoir of these pathogens. Therefore, oral hygiene in critically ill patients is an essential measure for the prevention of LRTIs, as recommended by both international and national guidelines.

Simple cleaning of the oral cavity using a toothbrush or oral swab, in addition to providing comfort and well-being to the patient, contributes to the prevention of LRTIs and other infections. A recent meta-analysis evaluating the impact of standardized toothbrushing on clinical outcomes showed that this care intervention was associated with a lower incidence of LRTIs and reduced mortality. On the other hand, an international clinical trial demonstrated that the implementation of an oral care bundle combined with the de-implementation of chlorhexidine for oral care was not associated with improved outcomes.

Based on the rationale supporting the benefits of implementing a standardized oral care, findings from previous studies, the conflicting literature regarding the effectiveness of oral care protocols that include the de-implementation of chlorhexidine on clinical outcomes in ICU patients, and the scarcity of data from developing countries such as Brazil, conducting a clinical trial is needed.

ELIGIBILITY:
Inclusion Criteria:

* All patients who receive mechanical ventilation in the participating intensive care units

Exclusion Criteria:

* Does not meet inclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4800 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2026-11-30 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
Ventilator free days | 28 days after enrollment
  Days alive and free from mechanical ventilation

SECONDARY OUTCOMES:
Intensive Care Unit all cause mortality | 15 months
  All cause mortality during intensive care unit stay
Hospital all cause mortality | 15 months
  All cause mortality during hospital stay
Ventilator associated pneumonia incidence | 15 months
  Defined as the number of ventilator associated pneumonia cases adjusted per ventilated-patients/days
Intensive care unit free days | 28 days after enrollment
  Days alive and free from intensive care unit
Hospital free days | 28 days after enrollment
  Days alive and free from hospital

CONTACTS AND LOCATIONS:
Overall Officials: Fernando Belissimo-Rodrigues, MD, PhD, Study Chair — Faculdade de Medicina de Ribeirão Preto da USP; Bruno M Tomazini, MD, Principal Investigator — Hospital do Coração (Hcor); Wanessa Belissimo-Rodrigues, PhD, Study Chair — Faculdade de Medicina de Ribeirão Preto da USP; Alexandre Biasi Cavalcanti, MD, PhD, Study Director — Hospital do Coração (Hcor)
Locations (6):
- Brazil (6):
  - Santa Casa de Misericordia de Passos, Passos, Minas Gerais
  - Hospital Municipal de Maringa, Maringá, Paraná
  - Hospital da Restauracao, Recife, Pernambuco
  - Hospital Santa Cruz, Santa Cruz, Rio Grande do Sul
  - Hospital Nereu Ramos, Florianópolis, Santa Catarina
  - Hospital Leo Orsi, Itapetininga, São Paulo

IPD SHARING:
Plan to Share IPD: Yes
Individual patient data (IPD) might be shared upon request and approval by the study committee after the study completion.
Supporting Information: Study Protocol, SAP
Time Frame: One year after study completion
Access Criteria: Individual patient data might be shared upon request and approval by the study committee after the study completion.

REFERENCES:
- [Result] Dale CM, Rose L, Carbone S, Pinto R, Smith OM, Burry L, Fan E, Amaral ACK, McCredie VA, Scales DC, Cuthbertson BH. Effect of oral chlorhexidine de-adoption and implementation of an oral care bundle on mortality for mechanically ventilated patients in the intensive care unit (CHORAL): a multi-center stepped wedge cluster-randomized controlled trial. Intensive Care Med. 2021 Nov;47(11):1295-1302. doi: 10.1007/s00134-021-06475-2. Epub 2021 Oct 5. PMID 34609548
- [Result] Price R, MacLennan G, Glen J; SuDDICU Collaboration. Selective digestive or oropharyngeal decontamination and topical oropharyngeal chlorhexidine for prevention of death in general intensive care: systematic review and network meta-analysis. BMJ. 2014 Mar 31;348:g2197. doi: 10.1136/bmj.g2197. PMID 24687313
- [Result] Bellissimo-Rodrigues WT, Menegueti MG, Gaspar GG, de Souza HCC, Auxiliadora-Martins M, Basile-Filho A, Martinez R, Bellissimo-Rodrigues F. Is it necessary to have a dentist within an intensive care unit team? Report of a randomised clinical trial. Int Dent J. 2018 Dec;68(6):420-427. doi: 10.1111/idj.12397. Epub 2018 May 18. PMID 29777534
- [Result] Bellissimo-Rodrigues F, Bellissimo-Rodrigues WT. Ventilator-associated pneumonia and oral health. Rev Soc Bras Med Trop. 2012 Oct;45(5):543-4. doi: 10.1590/s0037-86822012000500001. No abstract available. PMID 23152333
- [Result] Zhao T, Wu X, Zhang Q, Li C, Worthington HV, Hua F. Oral hygiene care for critically ill patients to prevent ventilator-associated pneumonia. Cochrane Database Syst Rev. 2020 Dec 24;12(12):CD008367. doi: 10.1002/14651858.CD008367.pub4. PMID 33368159
- [Result] Klompas M, Branson R, Cawcutt K, Crist M, Eichenwald EC, Greene LR, Lee G, Maragakis LL, Powell K, Priebe GP, Speck K, Yokoe DS, Berenholtz SM. Strategies to prevent ventilator-associated pneumonia, ventilator-associated events, and nonventilator hospital-acquired pneumonia in acute-care hospitals: 2022 Update. Infect Control Hosp Epidemiol. 2022 Jun;43(6):687-713. doi: 10.1017/ice.2022.88. Epub 2022 May 20. PMID 35589091
- [Result] Marino PJ, Wise MP, Smith A, Marchesi JR, Riggio MP, Lewis MAO, Williams DW. Community analysis of dental plaque and endotracheal tube biofilms from mechanically ventilated patients. J Crit Care. 2017 Jun;39:149-155. doi: 10.1016/j.jcrc.2017.02.020. Epub 2017 Feb 16. PMID 28259058
- [Result] van Nieuwenhoven CA, Buskens E, Bergmans DC, van Tiel FH, Ramsay G, Bonten MJ. Oral decontamination is cost-saving in the prevention of ventilator-associated pneumonia in intensive care units. Crit Care Med. 2004 Jan;32(1):126-30. doi: 10.1097/01.CCM.0000104111.61317.4B. PMID 14707570
- [Result] Magill SS, Edwards JR, Bamberg W, Beldavs ZG, Dumyati G, Kainer MA, Lynfield R, Maloney M, McAllister-Hollod L, Nadle J, Ray SM, Thompson DL, Wilson LE, Fridkin SK; Emerging Infections Program Healthcare-Associated Infections and Antimicrobial Use Prevalence Survey Team. Multistate point-prevalence survey of health care-associated infections. N Engl J Med. 2014 Mar 27;370(13):1198-208. doi: 10.1056/NEJMoa1306801. PMID 24670166
- [Result] Dasta JF, McLaughlin TP, Mody SH, Piech CT. Daily cost of an intensive care unit day: the contribution of mechanical ventilation. Crit Care Med. 2005 Jun;33(6):1266-71. doi: 10.1097/01.ccm.0000164543.14619.00. PMID 15942342